CLINICAL TRIAL: NCT07064460
Title: Duke Customized Aortic Aneurysm Repair With Endovascular Stent-grafts - Duke CARES Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chandler Long, MD (Other)
Responsible Party: Sponsor-Investigator, Chandler Long, MD, Associate Professor of Surgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00116274
Record Dates: First submitted 2025-06-26; First posted 2025-07-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Aortic Disorders
Keywords: aortic disorders; endovascular grafts
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Physician Modified Endovascular Graft (Experimental): The participant's surgeon will modify a commercially available graft tailored to their anatomy for their surgery.
  Interventions: Device: Physician Modified Endovascular Graft

INTERVENTIONS:
Device: Physician Modified Endovascular Graft — The participant's surgeon will modify a commercially available graft tailored to their anatomy for their surgery. All components used to create the final device (PMEG), made specifically for each participant and tailored to their individual anatomy, are FDA-approved, although the final graft itself (the PMEG) is considered investigational.

SUMMARY:
The purpose of this study is to see if physician modified endovascular grafts (PMEG) can be used safely for the treatment of aortic disorders. The surgeon will modify a commercially available graft tailored to the participant's anatomy for surgery. The researchers will follow participants for 5 years, which will require regular visits to the clinic for follow-up imaging and follow-up blood tests.

DETAILED DESCRIPTION:
The primary objective of the clinical investigation Duke CARES Trial is to assess the use of physician-modification of commercially available, off-the-shelf, endovascular stent-grafts to treat juxtarenal, pararenal and paravisceral complex abdominal aneurysms or thoracoabdominal aneurysms in high-risk for open surgery subjects having appropriate anatomy. The primary intent of the study is to assess safety and efficacy of the device acutely (i.e., treatment success and technical success), at 30 days (i.e., the rate of major adverse events (MAE)) and at 6 months, 12 months and annually to 5 years (i.e., the proportion of treatment group subjects that achieve and maintain treatment success).

Additionally, the study will assess domains for improvement of patient selection criteria, device design, operative techniques, and follow-up regimens to benefit patients undergoing complex endovascular aneurysm repair

Main Study - Statistical Cohort Physician Modified Endovascular Grafts are indicated for endovascular repair of juxtarenal, pararenal, paravisceral and thoracoabdominal aneurysms, in high-risk for open surgery subjects having appropriate anatomy as defined in the eligibility section.

Non-statistical cohort Patients with life-threatening aortic disease who have no acceptable surgical or endovascular alternatives will be allowed to receive treatment under this IDE. Enrollment of these patients under the IDE permits systematic data collection and FDA oversight, while their separation from the primary study cohort preserves the integrity of the safety and effectiveness analyses. This approach provides a treatment option for critically ill patients by offering access to a potential therapeutic option within a regulated and monitored environment without compromising the scientific validity of the trial. The patients in this cohort will follow standard of care, which includes follow-up at 1 month, 6 months and then annually. Data collection and presentation in this cohort will be consistent with the primary study cohort; however, data from this cohort will not be included in the statistical analysis.

ELIGIBILITY:
MAIN COHORT

INCLUSION CRITERIA:

* A participant may be entered into the study if the participant has at least one of the following: An aneurysm with a maximum diameter of > 5.5 cm or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e, perpendicular to the centerline) measurements; Aneurysm with a history of growth > 0.5 cm in 6 months; Saccular aneurysm deemed at significant risk for rupture; Symptomatic aneurysm; Ruptured aneurysm

AND

* Extent of aorta to be treated: juxtarenal, pararenal that include 1 or 2 renal and/or accessory renal arteries, paravisceral that includes celiac artery and/or superior mesenteric artery, and/or thoracoabdominal
* High risk of morbidity and mortality with open surgical repair as defined by:

  a. Anatomic Criteria (Previous abdominal surgery; Previous thoracotomy; Previous aortic surgery) b. Physiologic Criteria (ASA Category III or higher; Age >70 years; Previous myocardial infarction, coronary artery disease, or coronary artery stent; Coronary stress test with a reversible perfusion defect; Congestive heart failure (CHF); Chronic obstructive pulmonary disease (COPD))
* Iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit
* Nonaneurysmal aortic segment proximal to the aneurysm (neck) with a minimum neck length of 25 mm (Diameter in the range of 18 mm - 42 mm; Angle less than 60o relative to the axis of the aneurysm; Angle less than 60o relative to the axis of the suprarenal aorta);

  * Minimum branch vessel diameter greater than 5 mm
  * Iliac artery distal fixation site greater than 20 mm in length and diameter in the range of 9 mm - 21 mm (for use of ZFEN)
  * Contralateral iliac artery distal fixation site greater than 20 mm in length and diameter in the range of 7.5 mm - 20 mm.
  * Age: ≥ 18 years old
  * Life expectancy: > 2 years

EXCLUSION CRITERIA:

GENERAL EXCLUSION CRITERIA:

* Able to be treated in accordance with the instructions for use with a currently marketed endovascular prosthesis
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent by subject or legal representative
* Pregnant or breastfeeding
* Prefers to receive treatment at another hospital with access to a non-physician modified endovascular prosthesis
* Refusal of blood transfusions for religious or personal reasons
* Participation in another investigational clinical or device trial, with the exception of another investigational endovascular stent-graft protocol or percutaneous aortic valve protocol, not encompassed by the IDE protocol and performed remotely from the fenestrated procedure (> 30 days). Examples include remote (>30 days) participation in a thoracic, abdominal or iliac branch device trial, or participation in a percutaneous aortic valve trial.
* Mycotic aneurysm or evidence of active systemic infection

MEDICAL EXCLUSION CRITERIA:

* Known sensitivities or allergies to the materials of construction of the devices, including nitinol (nickel, titanium), polyester, polypropylene, gold, stainless steel, and/or solder (tin, silver).
* Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
* Uncorrectable coagulopathy
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment

  • Morbid obesity (BMI ≥ 40 or BMI 30-39.9 with comorbidities)
* Major surgical or interventional procedure unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
* Baseline creatinine greater than 2.0 mg/dL
* History of connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome)
* Deemed a high risk due to significant comorbidities, adjudicated by severity according to the Society for Vascular Surgery reporting standards for endovascular aortic repair involving the renal-mesenteric arteries

ANATOMICAL EXCLUSION CRITERIA:

* Thrombus or excessive calcification within the neck of the aneurysm
* Presence of significant thrombus and/or excessive calcification within the intended proximal or distal seal zone of the aneurysm.
* Branch stenosis > 75% (if left untreated)
* Anatomy that would not allow maintenance of at least one patent hypogastric artery

  * Inadequate femoral or iliac access to accommodate the required delivery systems.
  * Requirement for iliac conduit in cases of inadequate femoral/iliac access
  * Absence of a suitable non-aneurysmal segment of distal thoracic aorta and significant aortic tortuosity.
  * Target vessel anatomy not compatible with fenestrated or branched stent graft incorporation, including vessels with severe stenosis, tortuosity and/or insufficient size to accommodate stent graft placement.
  * Early target vessel bifurcation precluding safe or effective stent graft placement.
  * Unsuitable iliac artery fixation site and/or anatomy for iliac limb extension or iliac branch device placement, as defined by the device instructions for use

Note: Patients with life-threatening aortic disease who have no acceptable surgical or endovascular alternatives will be allowed to receive treatment under this IDE in the non-statistical cohort

Non-statistical Cohort

This cohort will include patients who meet the inclusion criteria and meet any of the above exclusion criteria* with the exception of the following:

* Able to be treated in accordance with the instructions for use with a currently marketed endovascular prosthesis
* Subject prefers to receive treatment at another hospital with access to a custom-made endovascular prosthesis
* Refusal to give informed consent by the subject or legal representative. Note: Inability to consent prior to surgery will not be exclusionary if it is for life-saving measures.
* Known sensitivities or allergies to the materials of construction of the devices will be allowed in a life-threatening situation where the patient would not survive open surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2030-12-11 (Estimated); Study Completion 2031-12-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse events (MAE) | 30 days, or during hospitalization if this exceeds 30 days
  The primary safety endpoint is freedom from major adverse events (MAE) at 30 days or during hospitalization if this exceeds 30 days.
  MAE include death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, stroke, and estimated procedural blood loss > 1000 cc.
Proportion of study participants with treatment success | 1 year
  Treatment success requires all the following criteria to be met:
  * Technical success
  * Absence of death from the initial procedure, secondary intervention, or aorta-related cause
  * Absence of persistent type I or type III endoleak
  * Absence of aneurysm sac expansion >5 mm
  * Absence of device migration >10 mm
  * Absence of failure due to device integrity issues
  * Absence of aneurysm rupture
  * Absence of conversion to open surgical repair
  * Device infection or thrombosis

SECONDARY OUTCOMES:
Technical success | Within 24 hours
  Technical success - defined as the successful introduction, deployment and withdrawal of the device, in the absence of surgical conversion or mortality, absence of Type I and III endoleak, absence of branch occlusion ensuring unimpeded flow to the branch vessel(s) intended for preservation or absence of graft limb obstruction.
Incidence of death | 30 days
Incidence of bowel ischemia | 30 days
Incidence of myocardial infarction | 30 days
Incidence of paraplegia | 30 days
Incidence of renal failure | 30 days
Incidence of respiratory failure | 30 days
Incidence of stroke | 30 days
Estimated procedural blood loss > 1000 cc | During procedure
Incidence of paraparesis | 30 days
Proportion of study participants with treatment success | 30 days, 6 months, 2 years, 3 years, 4 years, and 5 years
  Treatment success requires all the following criteria to be met: • Technical success • Absence of death from the initial procedure, secondary intervention, or aorta-related cause • Absence of persistent type I or type III endoleak • Absence of aneurysm sac expansion >5 mm • Absence of device migration >10 mm • Absence of failure due to device integrity issues • Absence of aneurysm rupture • Absence of conversion to open surgical repair • Device infection or thrombosis
Proportion of participants who experience any of the specified events | 30 days, 6 months, 12 months, 2 years, 3 years, 4 years, and 5 years
  Events include:
  * Aneurysm enlargement
  * Aneurysm-related mortality
  * Aneurysm rupture
  * Conversion to open repair
  * Secondary intervention for:
    * Migration
    * Type I (a, b, c) endoleak (See definitions and Figure 1)
    * Type III (a, b, c) endoleak (See definitions and Figure 1)
    * Device integrity failure (e.g., fracture)
    * Patency-related events (i.e., device stenosis or occlusion and embolic events)
  * Renal failure
  * All-cause mortality
  * Endoleaks
  * Device integrity failure (e.g., fracture)
  * Patency -related events (i.e., endovascular graft or stent component stenosis or occlusion and embolic events)
  * Other device-related events

CONTACTS AND LOCATIONS:
Overall Officials: Chandler Long, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No